CLINICAL TRIAL: NCT02472808
Title: Diagnostic Utility of EBUS-TBNA Versus Conventional TBNA With Rapid on Site Evaluation in the Diagnosis of Sarcoidosis: a Randomised Study
Brief Title: A Trial to Compare Two Methods of Obtaining Tissue for Diagnosis of Sarcoidosis Namely the Conventional Method or the Ultrasound Guided Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Ashesh Dhungana, Senior Resident, Department of Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DM Thesis
Record Dates: First submitted 2015-06-07; First posted 2015-06-16 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- cTBNA without ROSE (Other): Patients who will undergo conventional TBNA without ROSE + Endobronchial biopsy + Transbronchial Lung Biopsy
  Interventions: Other: cTBNA without ROSE
- cTBNA with ROSE (Other): Patients who will undergo conventional TBNA with ROSE + Endobronchial biopsy + Transbronchial Lung Biopsy
  Interventions: Other: cTBNA with ROSE
- EBUS-TBNA without ROSE (Other): Patients who will undergo EBUS-TBNA without ROSE + Endobronchial biopsy + Transbronchial Lung Biopsy
  Interventions: Other: EBUS-TBNA without ROSE
- EBUS-TBNA with ROSE (Other): Patients who will undergo EBUS-TBNA with ROSE + Endobronchial biopsy + Transbronchial Lung Biopsy
  Interventions: Other: EBUS-TBNA with ROSE

INTERVENTIONS:
Other: cTBNA without ROSE — Patients will undergo conventional TBNA and endobronchial biopsy and transbronchial lung biopsy
  Arms: cTBNA without ROSE
Other: cTBNA with ROSE — Patients will undergo conventional TBNA with rapid on site evaluation of cytology smear and endobronchial biopsy and transbronchial lung biopsy
  Arms: cTBNA with ROSE
Other: EBUS-TBNA without ROSE — Patients will undergo EBUS-TBNA and endobronchial biopsy and transbronchial lung biopsy
  Arms: EBUS-TBNA without ROSE
Other: EBUS-TBNA with ROSE — Patients will undergo EBUS-TBNA with rapid onsite evaluation of cytology smear and endobronchial biopsy and transbronchial lung biopsy
  Arms: EBUS-TBNA with ROSE

SUMMARY:
This trial compares the yield of cTBNA (conventional Transbronchial Needle Aspiration) versus the EBUS-TBNA (Endobronchial Ultrasound guided TBNA) for obtaining cytology when they are combined with endobronchial biopsy and transbronchial lung biopsy and rapid onsite examination (ROSE) of the obtained smears in the diagnosis of suspected sarcoidosis patients visiting our hospital for evaluation of mediastinal lymphadenopathy.

DETAILED DESCRIPTION:
This study is investigator initiated, prospective, unblinded randomized study comparing conventional TBNA with EBUS-TBNA for obtaining tissue samples from mediastinal lymph nodes for the diagnosis of sarcoidosis when combined with transbronchial lung biopsy and endobronchial biopsy. It will be conducted on 80 consecutive patients with suspected sarcoidosis presenting to Department of Pulmonary Medicine and Sleep Disorders in AIIMS (All India Institute of Medical Sciences), New Delhi. This study will help to know whether EBUS (Endobronchial Ultrasound guided) or conventional TBNA is better for obtaining tissue samples from mediastinal lymph nodes for the diagnosis of sarcoidosis. It will also help to know the value of adding rapid onsite evaluation of the cytology smears to both the procedures. It will also help to determine the overall yield of different procedures when they are combined for obtaining tissue samples for a diagnosis of sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and suspected Stage 1 (mediastinal or hilar Lymphadenopathy (LAP)) or Stage 2 ( LAP and parenchymal abnormalities) sarcoidosis
* Significant mediastinal LAP (Short Axis Diameter more than 10mm)
* Lymph Node (LN) enlargement in station 4, 7, 10 or 11 and CT chest findings consistent with sarcoidosis.
* With or without supportive evidence of sarcoidosis - hypercalcemia, calciuria, raised ACE levels or restriction/obstruction on Pulmonary Function Tests (PFT).

Exclusion Criteria:

* Obvious other organ involvement with possibility to confirm granuloma with minimally invasive diagnostic procedure (Skin biopsy, superficial lymph nodes, Lofgren's Syndrome)
* Sarcoidosis Stage 3 and 4
* Mediastinal Nodes less than 10 mm in short axis diameter
* Absence of right paratracheal and subcarinal Lymph node enlargement more than 1 cm in short axis diameter
* Those who received empiric Steroid for >2 weeks in preceding 3 months
* Contraindication to bronchoscopy and TBNA (Coagulopathy, Hypoxemia)
* Unwilling to give consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Yield of Conventional TBNA vs EBUS TBNA with or without ROSE | 6 months
  Diagnostic Yield is defined as the number of patients with presence of non caseating granuloma on cytology smear divided by total number of sarcoidosis patient expressed as percentage

SECONDARY OUTCOMES:
Yield of EBUS-TBNA in Conventional TBNA with or without ROSE negative patients | 6 months
  Yield is defined as the number of patients with presence of non caseating granuloma on cytology smear divided by total number of sarcoidosis patient expressed as percentage
Sensitivity of conventional TBNA to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Sensitivity of conventional TBNA when combined with ROSE to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Sensitivity of EBUS-TBNA to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Sensitivity of EBUS-TBNA when combined with ROSE to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Specificity of conventional TBNA to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Specificity of conventional TBNA when combined with ROSE to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Specificity of EBUS-TBNA to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Specificity of EBUS-TBNA when combined with ROSE to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Positive predictive value of conventional TBNA to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Positive predictive value of conventional TBNA when combined with ROSE to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Positive predictive value of EBUS-TBNA to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Positive predictive value of EBUS-TBNA when combined with ROSE to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Negative predictive value of conventional TBNA in the diagnosis of Sarcoidosis | 6 months
Negative predictive value of conventional TBNA when combined with ROSE in the diagnosis of Sarcoidosis | 6 months
Negative predictive value of EBUS-TBNA in the diagnosis of Sarcoidosis | 6 months
Negative predictive value of EBUS-TBNA when combined with ROSE in the diagnosis of Sarcoidosis | 6 months

OTHER OUTCOMES:
Sensitivity of endobronchial biopsy to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Specificity of endobronchial biopsy to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Positive predictive value of endobronchial biopsy to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Negative predictive value of endobronchial biopsy in the diagnosis of Sarcoidosis | 6 months
Sensitivity of transbronchial lung biopsy to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Specificity of transbronchial lung biopsy to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Positive predictive value of transbronchial lung biopsy to detect Non Caseating Granuloma for the diagnosis of Sarcoidosis | 6 months
Negative predictive value of transbronchial lung biopsy in the diagnosis of Sarcoidosis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashesh Dhungana, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India